CLINICAL TRIAL: NCT03066960
Title: Long-term Efficacy of Radiofrequency Neurotomy for Chronic Zygapophysial (Facet) Joint Related Neck Pain
Brief Title: Radiofrequency Neurotomy for Chronic Facet Joint Related Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Gunnvald Kvarstein, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015/2194
Record Dates: First submitted 2017-02-20; First posted 2017-03-01 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain
Keywords: radiofrequency neurotomy; zygapophyseal joint
MeSH Terms: conditions — Neck Pain | interventions — Denervation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency neurotomy group (Active Comparator): Unilateral radiofrequency neurotomy of medial branches to the dorsal ramus at one or two cervical levels
  Interventions: Procedure: Radiofrequency neurotomy
- Sham group (Sham Comparator): Unilateral sham treatment of medial branches to the dorsal ramus at one or two cervical levels
  Interventions: Procedure: Sham treatment

INTERVENTIONS:
Procedure: Radiofrequency neurotomy — RF neurotomy represents a nerve destructive, coagulating technique affecting the conduction through all nerve fibers.
  Arms: Radiofrequency neurotomy group
Procedure: Sham treatment — Sham treatment represents no coagulation of the nerve and will not affect the nerve conduction.
  Arms: Sham group

SUMMARY:
This is a single-center, double blind, sham-controlled randomized trial (N: 34) to assess the long term efficacy of RF neurotomy of cervical medial branches. Patients with chronic unilateral neck pain who are found eligible and achieve ≥50% pain relief of two predictive and comparative test blocks will be included in the trial in a primary analysis. We will further test whether a strict selection of ≥80% pain relief better predicts efficacious RF neurotomy compared with a less strict selection of ≥50% to <80%. After 6 months sham-treated patients may also be offered active unblinded RF treatment. Demographic and clinical data will be recorded at baseline while primary and secondary outcome measurements are recollected after 1, 3, 6, 9 and 12 months. Primary outcome measurements include self-reported neck function (NDI) and pain relief after 6 months.

DETAILED DESCRIPTION:
Chronic neck pain represents a common health problem. The mechanisms appear to be multifactorial. Researchers have suggested a disturbed interplay between the deep neck muscles and facet joints. In Europe and the US radiofrequency neurotomy has become a common treatment. The evidence base, however, is still insufficient. Thus, a double blind, sham-controlled, randomized, single-center trial is carried out. Based on current data and a single center study design, 34 randomized participants, completing the trial, have shown adequate to obtain sufficient statistical power. To simplify the data collection a digital internet based program is used. Patients with chronic unilateral neck pain, referred to Oslo University Hospital or responding to public announcements, and not responding to non-interventional treatment will be screened. Those who are found eligible and achieve ≥50% pain relief after predictive and comparative test blocks, will be included in the study. We will further test whether a strict selection of ≥80% pain relief better predicts efficacious RF neurotomy compared with a less strict selection of ≥50% to <80%. After 6 months participants who received sham and still suffer from neck pain, will be offered unblinded RF neurotomy and additional 12 month unblinded follow up if the results support this treatment. Demographic and clinical data will be recorded at baseline. The primary and secondary outcome measurements are recollected after 1, 3, 6, 9 and 12 months. Primary outcome measurements include self-reported neck function (NDI) and pain relief after 6 months. Regression analyses will be used to identify how pain relief of two test blocks and pain catastrophizing predict response to RF neurotomy. If RF neurotomy is found superior to sham treatment, this may be implemented in the national treatment program for selected patients with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria

* Min 18 years and Maximum 80 years
* Read and understand Norwegian
* Stable neck pain >12 months, with or without unilateral headache
* Average of worst pain intensity last three days ≥ 4 out of maximum 10
* Neck Disability Index >15 points or > 30 percentage points.
* At least two predictive blocks ≥ 50% pain relief 30 to 60 minutes after lidocaine and 30 to 180 minutes after bupivacaine .

Exclusion Criteria:

* Serious cervical pathology (acute cervical disc herniation, radiculopathy, myelopathy, spinal anomalies and chronic widespread pain
* Opioid consumption > 50 morphine equivalents/day
* Ongoing litigation process and applying for disability insurance/benefits
* Serious psychiatric disorder (DSM-IV-TR) diagnosed at a psychiatric unit, including suicidal thoughts and somatization (from Hopkins Symptom Check List 25 ≥ 2.5)
* Ongoing addictive behavior ( diagnostic criteria in Statistical Manual, 4th Edition)
* Unstable medical condition (ASA 4, serious vascular disease like unstable angina)
* Bacterial infection
* Malignancy
* Chronic generalized pain
* Hypersensitive to contrast agents or local anesthetics
* Pregnancy
* Bleeding diathesis
* Previously radiofrequency neurotomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-14 (Estimated); Study Completion 2025-12-14 (Estimated)

PRIMARY OUTCOMES:
Change in neck function after RF neurotomy vs sham treatment | 6 months
  Two independent group comparison of change of Neck Disability Index scores -continuous variable 0-50)
Change in pain intensity (numeric pain scale) after RF neurotomy vs sham treatment | 6 months
  Two independent group comparison of change in pain intensity (triplicate values from three consecutive days on a numeric pain scale 0-10 which provides a continuous variable)

SECONDARY OUTCOMES:
Change in neck function after RF neurotomy vs sham treatment | 12 months
  Two independent group comparison of change of Neck Disability Index scores -continuous variable 0-50
Change in pain intensity (numeric pain scale) after RF neurotomy vs sham treatment | 1 month
  Two independent group comparison of change in pain intensity (triplicate values from three consecutive days on a numeric pain scale 0-10 which provides a continuous variable)
Change in pain intensity (numeric pain scale) after RF neurotomy vs sham treatment | 3 months
  Two independent group comparison of change in pain intensity (triplicate values from three consecutive days on a numeric pain scale 0-10 which provides a continuous variable)
Change in pain intensity (numeric pain scale) after RF neurotomy vs sham treatment | 9 months
  Two independent group comparison of change in pain intensity (triplicate values from three consecutive days on a numeric pain scale 0-10 which provides a continuous variable)
Change in pain intensity (numeric pain scale) after RF neurotomy vs sham treatment | 12 months
  Two independent group comparison of change in pain intensity (triplicate values from three consecutive days on a numeric pain scale 0-10 which provides a continuous variable)
Change in pain intensity (categorical pain scale) after RF neurotomy vs sham treatment | 1 month
  Two independent group comparison of change in pain intensity (categorical 6-point pain scale with the alternatives worse, unchanged, <50% reduced, ≥50% reduced, and pain free which provides a categorial variable)
Change in pain intensity (categorical pain scale) after RF neurotomy vs sham treatment | 3 months
  Two independent group comparison of change in pain intensity (categorical 6-point pain scale wth the alternatives worse, unchanged, <50% reduced, ≥50% reduced, and pain free which provides a categorial variable)
Change in pain intensity (categorical pain scale) after RF neurotomy vs sham treatment | 6 months
  Two independent group comparison of change in pain intensity (categorical 6-point pain scale wth the alternatives worse, unchanged, <50% reduced, ≥50% reduced, and pain free which provides a categorial variable)
Change in pain intensity (categorical pain scale) after RF neurotomy vs sham treatment | 9 months
  Two independent group comparison of change in pain intensity (categorical 6-point pain scale wth the alternatives worse, unchanged, <50% reduced, ≥50% reduced, and pain free which provides a categorial variable)
Change in pain intensity (categorical pain scale) after RF neurotomy vs sham treatment | 12 months
  Two independent group comparison of change in pain intensity (categorical 6-point pain scale wth the alternatives worse, unchanged, <50% reduced, ≥50% reduced, and pain free which provides a categorial variable)
Change in health related quality of life after RF neurotomy vs sham treatment | 6 months
  Two independent group comparison of change of EuroQuol-5-Dimensions Index scores (continuous variable from -0.59 to 1.00)
Change in health related quality of life after RF neurotomy vs sham treatment | 12 months
  Two independent group comparison of change of EuroQuol-5-Dimensions Index scores (continuous variable from -0.59 to 1.00)
Change in drug consumption after RF neurotomy vs sham treatment | 6 months
  Two independent group comparison of change of the numbers of analgesic drugs (continuous variable)
Change in drug consumption after RF neurotomy vs sham treatment | 12 months
  Two independent group comparison of change of the numbers of analgesic drugs (continuous variable)
Change in number of neck/pain treatments after RF neurotomy vs sham treatment | 6 months
  Two independent group comparison of change of the numbers of neck/pain treatments (continuous variable)
How highly positive response to test block influences neck function after RF treatment | 6 months
  Regression analysis on how ≥80% pain relief (independent categorical variable) predicts >15% reduction of Neck disability Score (categorical variable) after RF neurotomy
How moderately positive response to test block influences neck function after RF treatment | 6 months
  Regression analysis on how ≥50% and <80% pain relief (independent categorical variable) predicts >15% reduction of Neck disability Score (categorical variable) after RF neurotomy
How highly positive response to test block influences 30% pain relief after RF treatment | 6 months
  Regression analysis on how ≥80% pain relief (independent categorical variable) predicts >30% reduction in pain intensity (categorical variable) after RF neurotomy
How moderately positive response to test block influences 30% pain relief after RF treatment | 6 months
  Regression analysis on how ≥50% and <80% pain relief (independent categorical variable) predicts >30% reduction in pain intensity (categorical variable) after RF neurotomy
How highly positive response to test block influences 50% pain relief after RF treatment | 6 months
  Regression analysis on how ≥80% pain relief (independent categorical variable) predicts >50% reduction in pain intensity (categorical variable) after RF neurotomy
How moderately positive response to test block influences 50% pain relief after RF treatment | 6 months
  Regression analysis on how ≥50 and <80% pain relief (independent categorical variable) predicts >50% reduction in pain intensity (categorical variable) after RF neurotomy
How catastrophizing influences neck function after RF treatment. | 6 months
  Regression analysis on how Pain Catastrophizing Scale score ≥30 (independent categorical variable) predict ≥ 15% reduction of Neck Disability Score (categorical variable) after RF neurotomy vs Pain Catastrophizing Scale score < 30
How catastrophizing influences pain relief after RF treatment. | 6 months
  Regression analysis on how Pain Catastrophizing Scale scores ≥30 (independent categorical variable) predict >30% reduction in pain intensity (categorical variable) after RF neurotomy vs Pain Catastrophizing Scale scores < 30
Change in mental distress after RF neurotomy vs sham treatment. | 6 months
  Two independent group comparison of change in Hopkin Symptom Check List (HSCL 25) sumscore which is a continuous variable on anxiety and depressive symptoms, ranging from 1 (normal) to 4 (worse)
Change in mental distress after RF neurotomy vs sham treatment. | 12 months
  Two independent group comparison of change in Hopkin Symptom Check List (HSCL 25) sumscore which is a continuous variable on anxiety and depressive symptoms, ranging from 1 (normal) to 4 (worse)
Change in sleep disturbances after RF neurotomy vs sham treatment. | 6 months
  Two independent group comparison of change in sleep. Sleep Subscale in Neck Disability Index part 7. A continuous variable based on a 6 point scale ranging from 0 to 6 where 0 is no problem and 6 i severe insomnia.
Change in sleep disturbances after RF neurotomy vs sham treatment. | 12 months
  Two independent group comparison of change in sleep. Sleep Subscale in Neck Disability Index part 7. A continuous variable based on a 6 point scale ranging from 0 to 6 where 0 is no problem and 6 i severe insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnvald Kvarstein, Dr. Med, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Department for Pain and Complex Disorders, Trondheim, Torgarden
  - Department of Pain Management and Research Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data Sharing Plan. In accordance with the general data sharing policy at OUH, the deidentified, individual data can be made available for external researchers from 9 months to 5 years after publication. However, to get access the researchers need to provide a methodologically sound proposal in accordance with the institutional guidelines and sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 9 months to 5 years after publication
Access Criteria: To get access the researchers need to provide a methodologically sound proposal in accordance with the institutional guidelines and sign a data access agreement.